CLINICAL TRIAL: NCT06177769
Title: Comparison of Efficacy and Complications of Three Supraglottic Airway Devices in Endobronchial Ultrasonographic Transbronchial Needle Aspiration Anesthesia
Brief Title: Comparison of Supraglottic Airway Devices in EBUS
Acronym: SAD-EBUS
Status: Completed | Type: Observational
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Derya Guzelkaya, Dr, Ankara Etlik City Hospital
Other Study IDs: SAD-EBUS Derya
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Airway Management; Lung Diseases
Keywords: Airway management; Lung diseases
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Group I: Airway is secured with LMA classic
  Interventions: Device: LMA classic
- Group II: Airway is secured with LMA proseal
  Interventions: Device: LMA Proseal
- Group III: Airway is secured with I-gel
  Interventions: Device: I-gel

INTERVENTIONS:
Device: LMA classic — Airway is secured with LMA clasic
  Groups: Group I
Device: LMA Proseal — Airway is secured with LMA proseal
  Groups: Group II
Device: I-gel — Airway is secured with I-gel
  Groups: Group III

SUMMARY:
Supraglottic airway devices (SAD) provide ventilation of patients requiring respiratory support without tracheal intubation. Therefore, SAD is used to maintain airway during anesthesia in surgeries that do not require intubation. The classical laryngeal mask (cLMA, Intavent Direct, Maidenhead, UK) is an SAD that is available as a more advanced airway method than mask ventilation and a less invasive method than endotracheal intubation. It is used by placing it over the glottis at the level of the larynx and inflating the cuff. The Proseal laryngeal mask (LMA-Proseal™, PLMA, Intavent Orthofix, Maidenhead, UK) is the first supraglottic airway device that is suitable for reuse and includes a gastric drainage channel. I-gel™ (Intersurgical Ltd, Wokingham, UK) is a second-generation laryngeal mask with a soft, gel-like thermoplastic elastomer distal end and no inflatable cuff, designed not to compress the anatomical structures of the larynx and pharynx.

Endobronchial ultrasound (EBUS)-guided transbronchial needle aspiration (TBNA) has become one of the most important invasive diagnostic procedures for pulmonologists and thoracic surgeons. It is a safe and effective technique for sampling hilar and mediastinal lymph nodes and masses. It is currently accepted as the first choice for histological sampling of the mediastinum in lung cancer staging.

The use of SAD to secure the airway in patients undergoing EBUS-TBNA has the advantages of being less invasive than endotracheal intubation and providing better surgical field access.

Classical LMA, proseal LMA and I-gel are routinely used airway methods during EBUS-TBNA procedure.

The aim of this study is to compare the routinely used SADs in anesthesia management in patients undergoing endobronchial ultrasonography-guided transbronchial needle aspiration in terms of intraoperative efficacy and postoperative complications.

DETAILED DESCRIPTION:
The parameters to be recorded are: demographic characteristics of the patients, hemodynamic data during and after the procedure, ventilation variables (tidal volume, airway pressures, leak volume), the number of attempts to place the SAD, the need for intubation, the presence of sore throat, nausea and vomiting after the procedure. In addition, the operator performing the procedure will be asked to evaluate the convenience of the procedure.

ELIGIBILITY:
Inclusion Criteria:

* adults ageing 18-80 years
* patients in ASA phyical class
* patients undergoing Endobronchial ultrasound guided transbronchial needle aspiration

Exclusion Criteria:

* patients undergoing emergent procedure
* pediatric patients
* patients having upper airway pathology
* patients in risk of aspiration

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing Endobronchial ultrasound guided transbronchial needle aspiration
Sampling Method: Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Quality of fiberoptic view | 3 minutes after anesthesia induction
  The operator will score the view of the glottic opening according to the Cormack Lehanne score

SECONDARY OUTCOMES:
Ease of passage through glottic opening | 3 minutes after anesthesia induction
  The operator will score theEase of passage through glottic opening according to a Likert scale
Ease of SAD insertion | 2 minutes after anesthesia induction
  The anesthetist will score the ease of SAD insertion a 5 point scale
Complications | 1 minute after extubation
  Airway trauma as indicated with blood stain on SAD or visible bleeding in the airway

CONTACTS AND LOCATIONS:
Overall Officials: Derya Güzelkaya, Dr, Principal Investigator — Ankara Etlik City Hospital
Locations (1):
- Etlik City Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Maitra S, Baidya DK, Arora MK, Bhattacharjee S, Khanna P. Laryngeal mask airway ProSeal provides higher oropharyngeal leak pressure than i-gel in adult patients under general anesthesia: a meta-analysis. J Clin Anesth. 2016 Sep;33:298-305. doi: 10.1016/j.jclinane.2016.04.020. Epub 2016 May 18. PMID 27555181
- [Background] Goel MK, Kumar A, Maitra G, Singh B, Ahlawat S, Jain P, Garg N, Verma RK. Safety and diagnostic yield of transbronchial lung cryobiopsy by flexible bronchoscopy using laryngeal mask airway in diffuse and localized peripheral lung diseases: A single-center retrospective analysis of 326 cases. Lung India. 2021 Mar-Apr;38(2):109-116. doi: 10.4103/lungindia.lungindia_220_20. PMID 33687002